CLINICAL TRIAL: NCT05911867
Title: The Combined Effect of Mulligan and Muscle Energy Techniques on Shoulder Kinematics and Postural Changes After Breast Cancer Surgery With Axillary Dissection: A Prospective, Randomized, Controlled Clinical Trial
Brief Title: Muscle Energy Technique and Mulligan's Mobilization in Breast Cancer Surgery Patients
Acronym: MWMMET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hany Mohamed Ibrahim Elgohary, Professor Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F.P.T2207005
Record Dates: First submitted 2023-06-11; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Mobility Limitation; Muscle Relaxation; Kinematics; Postural; Defect; Breast Cancer
MeSH Terms: conditions — Mobility Limitation; Breast Neoplasms | interventions — Movement

STUDY DESIGN:
Intervention Model Description: controlled, single-blinded, and randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: both participants and outcome assessors are blind for groups allocation and treatment modalities
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- combination of mobilization with movement and muscle energy techniques (Experimental): Mulligan technique (MWM) involves the therapist using a belt around the humeral head to guide appropriate gliding while the patient moves their shoulder actively through the range. The therapist applies pressure to the scapula in a counter direction.
  Regarding the cervical spine, the second technique, Cervical Self-Natural Apophyseal Glides (SNAG), involves the therapist standing behind the patient and applying force to the spinous process of each vertebra using a thumb-over-thumb technique.
  The examiner passively abducts the arm in the horizontal plane until the first barrier to motion by applying pressure to the distal humerus. This passive stretch will be held for three seconds.
  Interventions: Other: combination of mobilization with movement and muscle energy techniques
- mobilization with movement (Active Comparator): Regarding the shoulder joint, the Mulligan technique (MWM) involves the therapist using a belt around the humeral head to guide appropriate gliding while the patient moves their shoulder actively through the range. The therapist applies pressure to the scapula in a counter direction. This technique is usually performed for five sets of five repetitions with one minute of rest between sets in a sitting position.
  Regarding the cervical spine, the second technique, Cervical Self-Natural Apophyseal Glides (SNAG), involves the therapist standing behind the patient and applying force to the spinous process of each vertebra using a thumb-over-thumb technique. The patient actively performs repeated flexion or extension of their neck, returning back to the neutral position.
  Interventions: Other: mobilization with movement
- muscle energy techniques (Active Comparator): The examiner passively abduct the arm in the horizontal plane until the first barrier to motion by applying pressure to the distal humerus. This passive stretch will be held for three seconds. The examiner then instruct the participant to attempt to horizontally adduct the test arm at 25% of their maximal effort while the examiner applies manual resistance at the distal humerus to create an isometric contraction lasting five seconds. The participant then actively abduct the arm in the horizontal plane for a three-second active-assisted stretch.
  Interventions: Other: muscle energy techniques Interventions:

INTERVENTIONS:
Other: combination of mobilization with movement and muscle energy techniques — The examiner passively abducts the arm in the horizontal plane until the first barrier to motion by applying pressure to the distal humerus. The participant then actively abduct the arm in the horizontal plane for a three-second active-assisted stretch.
  Regarding the cervical spine, the second technique, Cervical Self-Natural Apophyseal Glides (SNAG), involves the therapist standing behind the patient and applying force to the spinous process of each vertebra using a thumb-over-thumb technique. The patient actively performs repeated flexion or extension of their neck, returning back to the neutral position. The passive gliding is maintained in the anterosuperior direction along the facet joint line while flexing or extending the neck throughout the range.
  Other Names: MWM
  Arms: combination of mobilization with movement and muscle energy techniques
Other: muscle energy techniques Interventions: — The examiner passively abduct the arm in the horizontal plane until the first barrier to motion by applying pressure to the distal humerus. This passive stretch will be held for three seconds. The examiner then instruct the participant to attempt to horizontally adduct the test arm at 25% of their maximal effort while the examiner applied manual resistance at the distal humerus to create an isometric contraction lasting five seconds. The participant then actively abduct the arm in the horizontal plane for a three-second active-assisted stretch.
  Other Names: MET
  Arms: muscle energy techniques
Other: mobilization with movement — Regarding the cervical spine, the second technique, Cervical Self-Natural Apophyseal Glides (SNAG), involves the therapist standing behind the patient and applying force to the spinous process of each vertebra using a thumb-over-thumb technique. The patient actively performs repeated flexion or extension of their neck, returning back to the neutral position. The passive gliding is maintained in the anterosuperior direction along the facet joint line while flexing or extending the neck throughout the range.
  Arms: mobilization with movement

SUMMARY:
A recent study aimed to examine the combined effect of Mulligan and muscle energy techniques on postural changes and shoulder kinematics among women who had undergone breast cancer surgery with axillary dissection.

DETAILED DESCRIPTION:
90 female patients who had undergone breast cancer surgery with axillary dissection were recruited and randomly assigned to three groups. Group A received Mulligan and muscle energy technique, group B received Mulligan technique only, and group C received muscle energy technique. The study measured shoulder kinematics and postural changes using a digital inclinometer for range of motion, PAS/SAPO for cervical angle, and the horizontal alignment of acromions and quick DASH for upper extremity activities. Outcome measurements were taken at three different time points: baseline, six weeks post-intervention, and eight weeks after the intervention during a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* female
* between 50 and 65 years
* limited shoulder range of motion

Exclusion Criteria:

* having metastases
* lymphedema
* traumatic or musculoskeletal disorders affecting the arm
* not taking anticoagulants
* not having undergone bilateral breast cancer surgery
* not having a locoregional recurrence
* not having vascular disorders in the affected arm

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
digital inclinometer | 6 weeks
  ). This tool is recognized as valid and reliable for this purpose and requires the patient to move their affected shoulder in various directions while keeping their feet fixed in place

SECONDARY OUTCOMES:
Postural Assessment Software (PAS/SAPO) | 6 weeks
  The women participants were positioned in a comfortable stance, and anatomical markers will be attached to specific points such as the tragus and both acromions. Their photographs will be captured and later analyzed using the PAS/SAPO software to record the cervical angle and horizontal alignment of the acromions. A forward head position was identified by an angle less than 50°. This method has been demonstrated to be reliable and valid for identifying forward head positions

OTHER OUTCOMES:
Quick DASH scale | 6 weeks
  The Arabic version of the Quick-DASH questionnaire includes 11 items, which inquire about the patient's difficulty in performing physical activities related to the upper extremity, the severity of pain and tingling, and the impact of the problem on social activities, work, and sleep. Each item includes five response options, ranging from no difficulty to being unable to perform the activity. If at least 10 items are answered, their responses are added to create a raw score, which is then transformed to a 0-100 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Hany M Elgohary, Principal Investigator — Delta University for Science and Technology, Gamasa, Coastal Road
Locations (1):
- Hany Mohamed Elgohary, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
i have no intent to share results

REFERENCES:
- [Background] Elgohary HM, Eladl HM, Soliman AH, Soliman ES. Effects of Ultrasound, Laser and Exercises on Temporomandibular Joint Pain and Trismus Following Head and Neck Cancer. Ann Rehabil Med. 2018 Dec;42(6):846-853. doi: 10.5535/arm.2018.42.6.846. Epub 2018 Dec 28. PMID 30613078